CLINICAL TRIAL: NCT05457088
Title: The Effect of High Protein on Body Composition and Markers of Sarcopenia in Patients With Type 2 Diabetes Mellitus
Brief Title: High Protein Effect on Body Composition and Sarcopenia Markers in Older Patients With Type 2 Diabetes Mellitus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National and Kapodistrian University of Athens (Other)
Collaborators: Harokopio University (Other)
Responsible Party: Principal Investigator, Vassilis Paschalis, Professor, National and Kapodistrian University of Athens
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 1288/03-07-2021
Record Dates: First submitted 2022-07-08; First posted 2022-07-13 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Type2 Diabetes Mellitus
Keywords: older adults; dietary protein; nutrition intervention; sarcopenia; performance; oxidative stress; inflammation; biochemical profile
MeSH Terms: conditions — Sarcopenia; Inflammation

STUDY DESIGN:
Intervention Model Description: 1st group will receive a dietary plan having dietary protein of 1.5gr/kg/day.2nd group will receive a dietary plan having dietary protein of 0.8gr/kg/day.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): Dietary intervention with protein intake 1.5 gr/kg/day
  Interventions: Other: 1.5 protein
- control group (Experimental): Dietary intervention with protein intake 0.8 gr/kg/day
  Interventions: Other: 0.8 protein

INTERVENTIONS:
Other: 1.5 protein — dietary plan having dietary protein of 1.5 gr/kg/day
  Arms: intervention group
Other: 0.8 protein — dietary plan having dietary protein of 0.8 gr/kg/day
  Arms: control group

SUMMARY:
This study will investigate the impact of dietary protein intake on progressive muscle loss and functionality (sarcopenia) in older adults with type 2 diabetes mellitus. Sarcopenia is known to have a bidirectional interaction with type 2 diabetes mellitus. Therefore in order to address this bidirectional complication we suggest that an increased intake of dietary protein at 1.5 gr/kg/day (current official recommendation is 0.8 gr/kg/day) could help to treat the sarcopenia, which in turn will help to ameliorate the type 2 diabetes mellitus progression.

ELIGIBILITY:
Inclusion Criteria:

* must have been diagnosed with type 2 diabetes mellitus during the last 5 years
* must have BMI 18.5-24.9

Exclusion Criteria:

* receive dietary supplements
* extreme dietary habits
* chronic inflammation disease
* cancer
* autoimmune disease

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-10-31 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
skeletal muscle mass index | Week 0, week 12
  Change from baseline in skeletal muscle mass index and will be assessed by dual energy x-ray absorptiometry ((leg lean mass+arm lean mass)/height^2)
calf circumference | Week 0, week 6, week 12
  Change from baseline in calf circumference and will be assessed by measuring tape
handgrip strength | Week 0, week 6, week 12
  Change from baseline in handgrip strength and will be assessed by handgrip dynamometer
Sit to stand test | Week 0, week 6, week 12
  Change from baseline in "Sit to stand" test which measures muscle functionality and will be assessed by chronometer
Timed up and go test | Week 0, week 6, week 12
  Change from baseline in "Timed up and go" test which measures muscle functionality and will be assessed by chronometer
10 meters walking test | Week 0, week 6, week 12
  Change from baseline in 10 meters walking test which measures muscle functionality and will be assessed by chronometer
blood glucose | Week 0, week 6, week 12
  Change from baseline in blood glucose and will be assessed by commercially available kit
Serum insulin | Week 0, week 6, week 12
  Change from baseline in serum insulin and will be assessed by commercially available kit
Glycosylated hemoglobin (HbA1) | Week 0, week 6, week 12
  Change from baseline in HbA1 and will be assessed by commercially available kit
C reactive protein | Week 0, week 6, week 12
  Change from baseline in C reactive protein and will be assessed by commercially available kit
Dietary intake of macro- and micro-nutrients | Week 0, week 3 , week 6, week 9, week 12
  Change from baseline in macro- and micro- nutrients and will be assessed with -3 day recall

SECONDARY OUTCOMES:
cholesterol level | Week 0, week 6, week 12
  Change from baseline in cholesterol level and will be assessed by commercially available kit
triglycerides level | Week 0, week 6, week 12
  Change from baseline in triglycerides level and will be assessed by commercially available kit
low-density lipoprotein (LDL) | Week 0, week 6, week 12
  Change from baseline in LDL and will be assessed by commercially available kit
high-density lipoprotein (HDL) | Week 0, week 6, week 12
  Change from baseline in HDL and will be assessed by commercially available kit
Enzymatic activity of glutathione peroxidase in plasma | Week 0, week 6, week 12
  Change from baseline in enzymatic activity of glutathione peroxidase in plasma and will be assessed by commercially available kit
Enzymatic activity of glutathione peroxidase in red blood cell lysate | Week 0, week 6, week 12
  Change from baseline in enzymatic activity of glutathione peroxidase in red blood cell lysate and will be assessed by commercially available kit
Enzymatic activity of superoxide dismutase in plasma | Week 0, week 6, week 12
  Change from baseline in superoxide dismutase in plasma and will be assessed by commercially available kit
Enzymatic activity of superoxide dismutase in red blood cell lysate | Week 0, week 6, week 12
  Change from baseline in superoxide dismutase in red blood cell lysate and will be assessed by commercially available kit
Protein carbonyls in plasma | Week 0, week 6, week 12
  Change from baseline in protein carbonyls in plasma and will be assessed by commercially available kit

CONTACTS AND LOCATIONS:
Locations (1):
- National and Kapodistrian University of Athens, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Result] Argyropoulou D, Geladas ND, Nomikos T, Paschalis V. Exercise and Nutrition Strategies for Combating Sarcopenia and Type 2 Diabetes Mellitus in Older Adults. J Funct Morphol Kinesiol. 2022 Jun 8;7(2):48. doi: 10.3390/jfmk7020048. PMID 35736019